CLINICAL TRIAL: NCT02521246
Title: Efficacy and Safety Evaluation of the New Association on Fixed Dose of Candesartan Cilexetil + Chlorthalidone (16mg + 12.5mg and 16mg + 25mg) Compared With HYZAAR® in Hypertension Control
Brief Title: Efficacy and Safety of Candesartan Associated With Chlorthalidone Versus Losartan Associated With Hydrochlorothiazide (Hyzaar®) in Essential Hypertension Control
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACEMS0315
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Essential Arterial Hypertension
MeSH Terms: interventions — candesartan; Chlorthalidone; hydrochlorothiazide, losartan drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test 1: Candesartan + Chlorthalidone (Experimental): The patients will take 1 tablet (Candesartan Cilexetil 16 mg + Chlorthalidone 12,5 mg) a day, in the morning.
  Interventions: Drug: Candesartan + Chlorthalidone
- Test 2: Candesartan + Chlorthalidone (Experimental): The patients will take 1 tablet (Candesartan Cilexetil 16 mg + Chlorthalidone 25 mg) a day, in the morning.
  Interventions: Drug: Candesartan + Chlorthalidone
- Comparator: Losartan+hydrochlorothiazide (Hyzaar®) (Active Comparator): The patients will take 1 tablet (Losartan 100 mg + Hydrochlorothiazide 25 mg) a day, in the morning.
  Interventions: Drug: Losartan+hydrochlorothiazide

INTERVENTIONS:
Drug: Candesartan + Chlorthalidone
  Arms: Test 1: Candesartan + Chlorthalidone
Drug: Candesartan + Chlorthalidone
  Arms: Test 2: Candesartan + Chlorthalidone
Drug: Losartan+hydrochlorothiazide
  Other Names: Hyzaar ®
  Arms: Comparator: Losartan+hydrochlorothiazide (Hyzaar®)

SUMMARY:
The purpose of this study is to evaluate the non-inferiority clinical efficacy of two different drug associations in the essential hypertension control.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent of the patient;
* Participants with decompensated essential hypertension, classified into stage 1 (with high or very high cardiovascular risk), stage 2 or stage 3 according to the Brazilian Society of Cardiology (2010), who are being treated with monotherapy.

Exclusion Criteria:

* Patients with any clinically significant disease that in the investigator opinion can not participate in the study;
* Secondary hypertension diagnosis or blood pressure above 190x100 mmHg in the screening/randomization visit;
* Morbid obesity or immunocompromised patients;
* Participants with greater than 10 mmHg difference in the measurements of systolic or diastolic blood pressure between the two arms;
* Participants who do not have the two upper limbs;
* Participants with important electrocardiographic changes;
* Creatinine clearance - less than 60 mL / min;
* History of hypertensive emergencies and cardiovascular and / or moderate to severe cerebrovascular events in the past 6 months;
* Microalbuminuria urine sample greater than 30 mg/g;
* Patients with history of hypersensitivity to any of the formula compounds;
* Pregnancy or risk of pregnancy and lactation patients;
* Participation in clinical trial in the year prior to this study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of essential hypertension control based on proportion of participants who achieve the therapeutic goal | 60 days

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences. | 9 weeks